CLINICAL TRIAL: NCT06382896
Title: A Clinical Study on the Effect of Oliceridine（TRV130） on Postoperative Rebound Pain and Early Rehabilitation Exercise After Knee Arthroscopy
Brief Title: Effect of Oliceridine on Rebound Pain
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Yang Bin, Principal Investigator, The First Affiliated Hospital of Xiamen University
Other Study IDs: FirstAHXiamenU-YB-2
Record Dates: First submitted 2024-04-15; First posted 2024-04-24 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Rebound Pain; Arthroscopic Knee Surgery; Oliceridine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing ambulatory arthroscopic knee surgery
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This was an observational study

SUMMARY:
The purpose of this clinical study was to identify the risk factors for postoperative pain outburst in patients undergoing arthroscopic knee surgery after Oliceridine and nerve block, and to evaluate the effect of oxeridine on early rehabilitation exercise in patients. A total of 320 patients undergoing arthroscopic knee arthroscopy under general anesthesia combined with femoral nerve block were selected to record the time and duration of postoperative pain outbreak, pain degree, age, gender, operation type, previous surgical history and other related risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old;2. Body mass index (BMI) 18-30kg /m2;3. American Society of Anesthesiologists (ASA) Grade I to II;4. Hospital stay >24h.

Exclusion Criteria:

1. Patients who cannot understand the numerical rating scale score and give feedback;2. Known allergy to the drug in the study;3. Infection of puncture site with nerve block;4. Oral analgesics for more than 2 weeks before surgery;5. Long-term use of glucocorticoids;6. Simultaneous surgery on both limbs;7. A psychopath;8. Severe compound trauma;9. Pregnant and lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General anesthesia combined with femoral nerve block was selected for knee arthroscopic day surgery
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time of onset of postoperative rebound pain | Within 48 hours after surgery
  The numerical rating scale was used
The duration of the rebound pain | Within 48 hours after surgery
  The numerical rating scale was used
The degree of the rebound pain | Within 48 hours after surgery
  The numerical rating scale was used
age | Within 48 hours after surgery
  Fill in the postoperative questionnaire
sex | Within 48 hours after surgery
  Fill in the postoperative questionnaire
Surgical procedure | Within 48 hours after surgery
  Fill in the postoperative questionnaire
Previous surgical history | Within 48 hours after surgery
  Fill in the postoperative questionnaire

SECONDARY OUTCOMES:
Movement recovery time | Within 7 days of surgery
  Fill in the postoperative questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China